CLINICAL TRIAL: NCT02476734
Title: A Pilot Study Using FDG-PET/CT Imaging as an Early Predictor of Disease Response in Lymphoma Subjects Receiving Redirected Autologous CART- 19 T-cell Immunotherapy
Brief Title: FDG-PET/CT Imaging as Early Predictor of DP
Status: Completed | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 12914
Record Dates: First submitted 2015-06-16; First posted 2015-06-19 (Estimated); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Lymphoma
Keywords: REDIRECTED AUTOLOGOUS CART- 19 T-CELL IMMUNOTHERAPY
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diffuse Large B-cell Lymphoma: There is no intervention. Will undergo baseline FDG-PET/CT to be performed within 6 weeks of infusion of CART-19 autologous T-cell therapy in a different study and then undergo repeat FDG-PET/CT at approximately 1 month after infusion. Infusion of CART-19 autologous T-cell therapy is not part of this study.
  Interventions: Other: There is no intervention
- Follicular Lymphoma: There is no intervention. Will undergo baseline FDG-PET/CT to be performed within 6 weeks of infusion of CART-19 autologous T-cell therapy in a different study and then undergo repeat FDG-PET/CT at approximately 1 month after infusion. Infusion of CART-19 autologous T-cell therapy is not part of this study.
  Interventions: Other: There is no intervention

INTERVENTIONS:
Other: There is no intervention — Subjects undergo FDG-PET CT scans in order to determine lesional FDG intake and changes in lesional FDG uptake.

SUMMARY:
In this study the investigators would like to describe FDG-PET/CT responses in patients who are receiving CART-19 immunotherapy for Follicular Lymphoma (FL), Diffuse Large B-cell Lymphoma (DLBCL), and Mantle Cell Lymphoma (MCL) as part of UPCC #13413. Subjects will undergo two FDG-PET/CTs. One performed within 6 weeks of CART-19 infusion and a repeat scan at about 1 month after infusion.

DETAILED DESCRIPTION:
In this study the investigators described FDG-PET/CT responses in patients who were receiving CART-19 immunotherapy for Follicular Lymphoma (FL), Diffuse Large B-cell Lymphoma (DLBCL), and Mantle Cell Lymphoma (MCL) as part of UPCC #13413. Subjects underwent two FDG-PET/CTs. One performed within 6 weeks of CART-19 infusion and a repeat scan at about 1 month after infusion.

ELIGIBILITY:
Inclusion Criteria:

* Subjects enrolled on the study UPCC 13413 Pilot Study Of Redirected Autologous T Cells Engineered To Contain Anti-Cd19 Attached To Tcr And 4-1bb Signaling Domains In Patients With Chemotherapy Resistant Or Refractory Cd19+ Lymphoma CART-19 autologous T-cell trial with relapsed or refractory DLBCL and FL. As this is a pilot study, we plan to enroll 4 subjects from the two disease types of interest.
* Subjects ≥ 18 years of age
* Subjects able to provide informed consent and agree to comply with study procedures

Exclusion Criteria:

* Subjects who are pregnant or lactating.
* Subjects will be co-enrolled in this study and UPCC 13413 and therefore must comply with the UPCC 13413 Pilot Study Of Redirected Autologous T Cells Engineered To Contain Anti-Cd19 Attached To Tcr And 4-1bb Signaling Domains In Patients With Chemotherapy Resistant Or Refractory Cd19+ Lymphoma requirements pertaining to pregnancy, lactation, conception and contraception use throughout their participation in both studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with DLBCL and FL treated on a phase I study with Autologous T cells
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2014-08; Primary Completion 2016-02 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Global objective tumor response measured from serial PET/CT scans | 1 month
  global objective tumor response measured from serial PET/CT scans as the change (absolute and relative (%)) in total metabolically active tumor volume (i.e., the total volume (in cc) of FDG-avid tumor throughout the body) between pre-treatment and post-treatment PET/CT scans.

CONTACTS AND LOCATIONS:
Overall Officials: Jakub Svoboda, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States